CLINICAL TRIAL: NCT04755582
Title: SMARTHEART Validation Study. A Study to Assess the Accuracy and Validate Novel Smartphone and Wearable ECG Devices in Cardiovascular Patients
Brief Title: SMARTHEART Validation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0693
Record Dates: First submitted 2021-02-05; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases
Keywords: wearable ecg; electrocardiogram
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the accuracy of novel smartphone or wearable ECG devices to a gold standard ECG in patients with normal and abnormal ECGs.

DETAILED DESCRIPTION:
Assess the effect of the following on the accuracy of the recorded ECG compared to a gold standard ECG:

* Posture or position of the patient
* Movement
* Amount of hair on the ECG site
* Skin condition (tone/dryness) Ability to detect a paced rhythm accurately A qualitative assessment of ECG devices, including the amount of artefact in the signal and ease of use of the device

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Must have an adequate understanding of written and spoken English
* Able (in the Investigators opinion) and willing to comply with study requirements.
* Must be over 18 years of age
* Must be deemed clinically stable by their direct care team.

Exclusion Criteria:

* Subjects who do not have an adequate understanding of written and spoken English
* Patients who are medically unstable, as defined by the patient's direct care team.
* Patients who are unable to give informed consent
* Patients who are deemed clinically unstable by their direct care team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from cardiology wards across the University Hospitals of Leicester trust.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of smartphone or wearable ECG devices compared to gold standard ECG devices | 2 hours
  To compare the accuracy of novel smartphone or wearable ECG devices to a gold standard ECG in patients with normal and abnormal ECGs.

SECONDARY OUTCOMES:
Assessing the effects on the ECG of: - Posture or position of the patient | 2 hours
  Assessment of changes to the ECG signal due to posture or position of the patient
Assessing the effects on the ECG of: • Movement | 2 hours
  Assessment of changes to the ECG signal due to movement of the patient
Assessing the effects on the ECG of: • Amount of hair on the ECG site | 12 months
  Assessment of changes to the ECG signal due to amount of hair on the site of ECG electrode positions
Assessing the effects on the ECG of: • Skin condition (tone/dryness) | 12 months
  Assessment of changes to the ECG signal due to different skin conditions on the site of ECG electrode positions
Ability to detect a paced rhythm accurately. | 2 hours
  Assessment of ability of ECG device to detect paced ECG complexes or pacing spikes
A qualitative assessment of ECG devices, including the amount of artefact in the signal and ease of use of the device. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: G. Andre Ng, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No